CLINICAL TRIAL: NCT06349148
Title: The Effects of Immunonutrition Therapy on the Nutritional Status, Immune Function, and Quality of Life of Locally Advanced Cervical Cancer Patients With Malnutrition: an Open-label Randomized Controlled Study
Brief Title: The Effects of Immunonutrition Therapy on Locally Advanced Cervical Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SHUANG ZHENG JIA, PhD (Other)
Responsible Party: Sponsor-Investigator, SHUANG ZHENG JIA, PhD, Attending Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NESTLE2022QN-0007
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancers
Keywords: Cervical cancer; Immunonutrition; Concurrent chemoradiotherapy; GLIM; Sarcopenia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immunonutrition (Experimental): enteral immunonutrition
  Interventions: Dietary Supplement: enteral immunonutrition
- standard nutrition (Active Comparator): standard oral enteral nutrition
  Interventions: Dietary Supplement: standard oral enteral nutrition

INTERVENTIONS:
Dietary Supplement: enteral immunonutrition — Patients in this group receives 2 bottles of immunonutrients per day (Impact, Nestlé, approximately 700 kcal).
  Arms: immunonutrition
Dietary Supplement: standard oral enteral nutrition — Patients in the control group receives isoenergetic standard oral enteral nutrition ( emulsion or Nutrison).
  Arms: standard nutrition

SUMMARY:
The goal of this open-label randomized control trial is to study the effect of immunonutrition in locally advanced cervical cancer (LACC) with standard concurrent chemoradiotherapy. LACC patients undergoing radical synchronous chemoradiotherapy will be randomized into the experimental group receiving enteral immunonutrition therapy and the control group receiving standard enteral nutrition support.The main purpose it aims to answer are:1）Can immunonutrition therapy improve patients' dose-limiting toxicity(DLT) and DLT-free survival? 2）Can immunonutrition therapy improve patients' nutritional status and quality of life?

DETAILED DESCRIPTION:
Malnutrition is one of the most common complications in patients with Locally Advanced Cervical Cancer (LACC) undergoing radical concurrent chemoradiotherapy (CCRT). Tumor patients often experience significant immune imbalance, metabolic abnormalities, and inflammatory responses. Immunonutrition therapy involves the use of specific immunonutrients such as polyunsaturated fatty acids, arginine, nucleotides, etc., to prevent and correct malnutrition in cancer patients, regulate immune function, alleviate harmful or excessive inflammatory responses, and thereby improve patients' clinical outcomes.

This study is an open-label randomized controlled trial, including patients with LACC who all receive radical radiotherapy. Using the Nutritional Risk Screening 2002 (NRS2002) at screening, patients identified as having nutritional risk are further assessed by nutritionists and physicians using the Patient-Generated Subjective Global Assessment (PG-SGA) score and modified Global leadership initiative on malnutrition (GLIM) criteria. Patients with moderate or severe malnutrition are randomly allocated into the enteral immunonutrition therapy group (experimental group) and the standard enteral nutrition support group (control group). The experimental group receives immunonutrients per day, while the control group receives isoenergetic standard oral enteral nutrition. Upon admission, all patients receive nutritional education from specialized nurses and consult with nutritionists, and nutritional support is provided during the concurrent chemoradiotherapy for a total of 5 weeks (W0-W5).GLIM score, quality of life score and peripheral blood inflammation and immune indicators were collected within 48 hours after admission (before treatment), W5, W8, and W20; CTCAE v 5.0 score was used for treatment side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Pathological histological diagnosis confirmed as cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma;
* Confirmed as Locally Advanced Cervical Cancer (LACC) based on gynecological examination and imaging assessment;
* Undergoing CCRT/RT treatment;
* Patients are conscious, able to communicate without barriers, and able to answer questions.
* diagnosed with malnutrition according to the GLIM criteria;

Exclusion Criteria:

* Patients who received neoadjuvant chemotherapy or immunotherapy before treatment;
* Patients with concomitant other malignant tumors or a history of malignant tumors;
* Patients with special pathological types of tumors such as cervical small cell carcinoma or neuroendocrine tumors;
* Patients staged as Ⅳb according to the International Federation of Gynecology and Obstetrics(FIGO) 2018 staging system;
* Patients with other severe chronic debilitating diseases, such as severe heart failure (New York Heart Association Class II-IV), severe liver damage (alanine aminotransferase ≥ 3 times the upper limit of normal), severe renal insufficiency (GFR < 30 ml/min*1.73 m²), etc.;
* Eastern Cooperative Oncology Group(ECOG) performance status ≥ 2;
* Presence of other contraindications to CCRT/RT.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 5-6 weeks
  Patients need to receive cisplatin treatment at 40 mg/m2 weekly for 5-6 weeks. During this period, any serious adverse reactions that lead to treatment interruption, delay, or chemotherapy dose reduction are defined as dose-limiting toxicities(DLT).
DLT-free survival | 5-6 weeks
  Time from start of treatment to onset of DLT

SECONDARY OUTCOMES:
compliance | 5-6 weeks
  the proportion of people who complete the prescribed treatment plan
Prevalence of malnutrition | 5-6 weeks, 3 months post-treatment
  assessed by GLIM criteria
Prevalence of sarcopenia | 5-6 weeks, 3 months post-treatment
  assessed by Skeletal muscle index(SMI) at the third lumbar vertebra(L3-SMI )calculated based on CT
QoL (Quality of life) | 5-6 weeks, 3 months post-treatment
  Quality of life measured by standardized EORTC quality of life questionnaire(QLQ)-C30
Objective response rate (ORR) | 3 months post-treatment
  evaluated by RECIST
laboratory tests | 5-6 weeks, 3 months post-treatment
  inflammation and immune-related indicators
2-year overall survival | 2 years
  the time from the start of treatment until the date of death from any cause
2-year progression-free survival | 2 years
  the date of the treatment to the date of disease progression or death from any cause in the absence of progression

CONTACTS AND LOCATIONS:
Overall Officials: SHUANGZHENG JIA, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No